CLINICAL TRIAL: NCT05850962
Title: Individualised Blood Pressure Targets Versus Standard Care Among Critically Ill Patients With Shock - A Multicentre Randomised Controlled Trial
Brief Title: Individualised Blood Pressure Targets Versus Standard Care Among Critically Ill Patients With Shock
Acronym: REACT-SHOCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rakshit Panwar (Other)
Responsible Party: Sponsor-Investigator, Rakshit Panwar, Conjoint Associate Professor, University of Newcastle, Australia
Organization: University of Newcastle, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: G2200761; ACTRN12623000044628 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2023-04-29; First posted 2023-05-09 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Critical Illness; Shock
Keywords: Relative hypotension
MeSH Terms: conditions — Critical Illness; Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard MAP target (No Intervention): The comparator or the control group will be comprised of patients assigned to standard care, where vasopressor support will be titrated to maintain a default MAP of 65 mmHg, unless the treating clinician considers a different MAP target as more appropriate.
- Individualised MAP target (Active Comparator): In the intervention arm, a patient's own pre-illness mean arterial pressure (MAP) would be targeted (range: 55-95 mmHg) during vasopressor support in ICU. The pre-illness MAP will be estimated from most recent pre-illness BP readings following a standardized method (Panwar et al,. Blood Press. 2017:1-9) and will be targeted for the duration of vasopressor therapy for up to a maximum of five days. The treating clinician can tailor these BP targets as deemed suitable for current clinical state. The type of vasopressor that will be used is at the discretion of the treating clinician.
  Study intervention will cease if a patient is considered well enough by the treating clinician for discharge out of ICU. If a patient is transported out of ICU for procedural intervention, then standard (non-study) treatment should be provided.
  Interventions: Other: Individualised MAP target

INTERVENTIONS:
Other: Individualised MAP target — The project will test an intervention that initially targets a patient's own pre-illness mean arterial pressure (MAP) during vasopressor support in ICU. The pre-illness MAP will be estimated from the most recent pre-illness BP readings recorded in medical records.
  Arms: Individualised MAP target

SUMMARY:
Aim The aim of the proposed RCT is to determine effectiveness of a strategy, where MAP (mean arterial blood pressure) targets during vasopressor therapy for shock in ICU are individualized based on patients' own pre-illness MAP that would be derived as an average of up to five most recent pre-illness blood pressure readings.

Hypothesis We hypothesize that targeting a patient's pre-illness MAP during management of shock can minimize the degree of MAP-deficit (a measure of relative hypotension), which may help reduce the risk of 14-day mortality and major adverse kidney events by day 14 in ICU.

Endpoints The primary endpoint will be the all-cause mortality rate at day 14. Secondary endpoints will be the time to death through day 14 and day 90, major adverse kidney events (MAKE-14), renal replacement therapy (RRT) free days until day 28, and 90-day all-cause mortality.

Significance To date no major RCT has tested this strategy among ICU patients with shock. This pivotal trial will provide evidence to fulfil a crucial knowledge gap regarding a common and a fundamental intervention in critical care.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients aged greater than or equal to 40 years
* The patient is deemed to be in shock, defined as clinician-initiated vasopressor/inotropic therapy AND supported by any of the following within the last 24 hours:

  * Lactate level greater than or equal to 2 mmol/l or base deficit greater than or equal to 3 mmol/l,
  * Urine output less than or equal to 0.5 ml/kg/h or <40 ml/h for 2 or more consecutive hours
  * Respiratory rate >22 per minute
  * Altered mentation (Glasgow Coma Score <14)

Exclusion Criteria:

* Patients who are moribund, or have documented not-for-resuscitation orders
* At least 24 hours have lapsed from the time of initiation of vasopressor or inotropic support
* Patients who are either receiving or are deemed to imminently need renal replacement therapy.
* Patients who already have an increase in serum creatinine of >350 µmol/l from baseline.
* End stage renal disease
* Patients where trauma is the main reason for the current ICU admission.
* Previously enrolled in the REACT Shock RCT
* Pregnancy, if known
* Active bleeding (clinical suspicion or >2 packed red blood cells within last 24 hours)
* Insufficient (less than two) pre-illness BP readings are available.
* Patients on extracorporeal support (such as extracorporeal membrane oxygenation, intra-aortic balloon pump, or ventricular assist device).
* Potential contraindications to either higher or lower BP targets (including but not limited to)

  * Cerebral perfusion pressure guided therapy e.g. intracranial hemorrhage or subarachnoid hemorrhage or traumatic brain injury
  * Abdominal perfusion pressure guided therapy
  * Aortic injury (e.g. dissection or post-operative)
  * Post cardiac surgery
  * Any other condition requiring higher or lower BP target specifically

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 14 days
  All deaths from randomisation to 14 days

SECONDARY OUTCOMES:
Time to death through day 14 | First 14 days of randomisation
Major Adverse Kidney Events | 14 days from randomisation
  Defined as a composite of death, new renal replacement therapy, or final serum creatinine level >= 200% of the latest preillness creatinine level, as assessed from patient medical records.
Renal replacement therapy free days until day 28 | 28 days from randomisation
Peak increase in serum creatinine levels | 28 days from randomisation
Time to death through day 90 | First 90 days of randomisation
Mortality | 90 days
  All deaths from randomisation to 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Medical Research Institute, Newcastle, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panwar R. Untreated Relative Hypotension Measured as Perfusion Pressure Deficit During Management of Shock and New-Onset Acute Kidney Injury-A Literature Review. Shock. 2018 May;49(5):497-507. doi: 10.1097/SHK.0000000000001033. PMID 29040214
- [Result] Panwar R, Tarvade S, Lanyon N, Saxena M, Bush D, Hardie M, Attia J, Bellomo R, Van Haren F; REACT Shock Study Investigators and Research Coordinators. Relative Hypotension and Adverse Kidney-related Outcomes among Critically Ill Patients with Shock. A Multicenter, Prospective Cohort Study. Am J Respir Crit Care Med. 2020 Nov 15;202(10):1407-1418. doi: 10.1164/rccm.201912-2316OC. PMID 32614244
- [Result] Panwar R, Van Haren F, Cazzola F, Nourse M, Brinkerhoff G, Quail A. Standard care versus individualized blood pressure targets among critically ill patients with shock: A multicenter feasibility and preliminary efficacy study. J Crit Care. 2022 Aug;70:154052. doi: 10.1016/j.jcrc.2022.154052. Epub 2022 May 5. PMID 35525132
- [Result] Panwar R, Lanyon N, Davies AR, Bailey M, Pilcher D, Bellomo R. Mean perfusion pressure deficit during the initial management of shock--an observational cohort study. J Crit Care. 2013 Oct;28(5):816-24. doi: 10.1016/j.jcrc.2013.05.009. Epub 2013 Jul 10. PMID 23849541
- [Result] Panwar R, Sullohern B, Shiel E, Alexis Brown C, Quail A. Validity of a protocol to estimate patients' pre-morbid basal blood pressure. Blood Press. 2018 Feb;27(1):10-18. doi: 10.1080/08037051.2017.1358055. Epub 2017 Jul 26. PMID 28745077
- [Derived] Panwar R, Gibberd A, Oldmeadow C, Tiruvoipati R, Aneman A, Kansal A; REACT SHOCK investigators. REACT SHOCK trial protocol and analysis plan-a multicenter randomised controlled trial comparing individualised blood pressure target versus standard blood pressure target among critically ill patients with shock. Trials. 2025 Oct 14;26(1):409. doi: 10.1186/s13063-025-09142-9. PMID 41088147